CLINICAL TRIAL: NCT02892760
Title: Clinical Algorithm for Post-Stroke Gait Training With C-Brace
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Otto Bock Healthcare Products GmbH (Industry)
Responsible Party: Principal Investigator, Gerard Francisco, Professor and Chairman of Physical Medicine and Rehabilitation, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-16-0031
Record Dates: First submitted 2016-08-02; First posted 2016-09-08 (Estimated); Results first posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Hemiparesis Due to Stroke; Hemiplegia Due to Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- with C-brace (Experimental): C-Brace is a micro-computer controlled brace that is worn on the leg to assist with walking.
  Interventions: Device: C-Brace

INTERVENTIONS:
Device: C-Brace — C-Brace is a micro-computer controlled brace that is worn on the leg to assist with walking.

SUMMARY:
The purpose of this study is to develop a clinical algorithmic-based evaluation and treatment approach for C-Brace for use by persons with hemiparesis or hemiplegia due to stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65 years
* Diagnosis of hemiparesis or hemiplegia following stroke
* Presence of abnormal walking pattern
* Poor knee control during stance phase
* Cognitive ability to (or care provider) manage daily charging of battery
* Cognitive ability to follow commands
* Hip flexor muscle strength grade 3 or greater or the ability to perform reciprocal gait using compensatory patterns

Exclusion Criteria:

* Weight > 275 lbs. (Includes body weight and weight of heaviest object carried)
* Less than 2° of ankle motion
* Severe spasticity of the quadriceps (MAS >3) and/or uncontrolled spasticity of the quadriceps
* Severe spasticity of other lower limb muscles (MAS >3)
* Fixed genuvalgum exceeding 10° beyond anatomic neutral valgum
* Any fixed genuvarum exceeding anatomic neutral varum.
* Hip or knee flexion contractures greater than 10°
* Presence of chronic obstructive pulmonary disease (COPD)
* Chronic heart failure - New York Heart Association (NYHA) stages 3 and 4

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Francisco, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- TIRR Research Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | With C-brace
Started | 17
Received Intervention | 15
Completed | 14
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for the 15 participants who received the intervention.
Arm/Group | With C-brace
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Gait Quality as Indicated by Joint Excursion as Assessed by Kinematic Analysis
Description: During the 10 Meter Walk Test (10MWT), infrared light emitting diode markers will be attached to bilateral lower extremities. The marker data will be recorded using the Northern Digital Inc (NDI) Optotrak Certus motion capture system. Marker data will be processed using custom Matlab program to determine lower extremity joint excursion. Joint excursion is the range of motion of a particular joint, and the range of motion is reported in degrees. After stroke, one side of the body is affected, and joint excursion for various joint angles (of hip, knee, and ankle) are reported for both sides of the body (affected side of body and unaffected side of body).
Time Frame: week 5
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | With C-brace
Number analyzed (Participants) | 11
degrees
  Affected Hip flexion-extension | 33.98 (10.03)
  Affected Hip abduction-adduction | 9.34 (3.04)
  Affected Hip internal-external rotation | 21.25 (14.45)
  Affected Knee flexion-extension | 34.51 (16.55)
  Affected Knee abduction-adduction | 7.72 (1.77)
  Affected Knee internal-external rotation | 16.26 (9.53)
  Affected Ankle flexion-extension | 13.51 (7.73)
  Affected Ankle abduction-adduction | 6.06 (4.33)
  Affected Ankle internal-external rotation | 8.36 (7.09)
  Unaffected Hip flexion-extension | 45.31 (10.21)
  Unaffected Hip abduction-adduction | 8.74 (3.11)
  Unaffected Hip internal-external rotation | 14.82 (6.41)
  Unaffected Knee flexion-extension | 53.71 (7.64)
  Unaffected Knee abduction-adduction | 10.30 (4.79)
  Unaffected Knee internal-external rotation | 11.83 (3.11)
  Unaffected Ankle flexion-extension | 21.83 (6.36)
  Unaffected Ankle abduction-adduction | 6.85 (1.75)
  Unaffected Ankle internal-external rotation | 12.64 (4.20)

2. Primary Outcome: Gait Quality as Indicated by Joint Excursion as Assessed by Kinematic Analysis
Description: During the 10 Meter Walk Test (10MWT), infrared light emitting diode markers will be attached to bilateral lower extremities. The marker data will be recorded using the NDI Optotrak Certus motion capture system. Marker data will be processed using custom Matlab program to determine lower extremity joint excursion. Joint excursion is the range of motion of a particular joint, and the range of motion is reported in degrees. After stroke, one side of the body is affected, and joint excursion for various joint angles (of hip, knee, and ankle) are reported for both sides of the body (affected side of body and unaffected side of body).
Time Frame: week 9
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | With C-brace
Number analyzed (Participants) | 11
degrees
  Affected Hip flexion-extension | 38.80 (11.26)
  Affected Hip abduction-adduction | 9.03 (3.55)
  Affected Hip internal-external rotation | 22.75 (15.71)
  Affected Knee flexion-extension | 34.93 (17.02)
  Affected Knee abduction-adduction | 7.92 (2.93)
  Affected Knee internal-external rotation | 16.18 (7.71)
  Affected Ankle flexion-extension | 15.91 (6.82)
  Affected Ankle abduction-adduction | 6.82 (5.51)
  Affected Ankle internal-external rotation | 7.55 (6.01)
  Unaffected Hip flexion-extension | 46.20 (10.79)
  Unaffected Hip abduction-adduction | 9.86 (3.34)
  Unaffected Hip internal-external rotation | 14.99 (5.25)
  Unaffected Knee flexion-extension | 55.55 (7.64)
  Unaffected Knee abduction-adduction | 12.06 (5.83)
  Unaffected Knee internal-external rotation | 12.78 (4.32)
  Unaffected Ankle flexion-extension | 21.88 (4.78)
  Unaffected Ankle abduction-adduction | 7.85 (2.17)
  Unaffected Ankle internal-external rotation | 13.16 (5.42)

3. Primary Outcome: Change in Muscle Function as Indicated by EMG Amplitude Assessed by Surface Electromyography (sEMG)
Description: Bipolar surface electrodes will be placed on the bilateral major leg muscles to record electromyography (1000Hz, Motion Labs 16-Channel EMG System). The EMG amplitude (in volts) will be calculated over the whole gait cycle during the 10 Meter Walk Test (10MWT), in which the participant walks 10 meters. After stroke, one side of the body is affected, and data for various muscles are reported for both sides of the body (affected side of body and unaffected side of body).
Time Frame: week 5
Measure: Mean (Standard Deviation); unit: volts
Arm/Group | With C-brace
Number analyzed (Participants) | 11
volts
  Affected Tibialis anterior | 0.2627 (0.0914)
  Affected Soleus | 0.2484 (0.0641)
  Affected Medial gastrocnemius | 0.2183 (0.1011)
  Affected Vastus medialis | 0.2211 (0.0837)
  Affected Rectus femoris | 0.2513 (0.0607)
  Affected Biceps femoris | 0.3136 (0.0723)
  Affected Semimembranous | 0.2184 (0.0734)
  Unaffected Tibialis anterior | 0.2791 (0.0595)
  Unaffected Soleus | 0.3095 (0.0574)
  Unaffected Medial gastrocnemius | 0.2322 (0.0898)
  Unaffected Vastus medialis | 0.2508 (0.0827)
  Unaffected Rectus femoris | 0.2827 (0.0873)
  Unaffected Biceps femoris | 0.2654 (0.0912)
  Unaffected Semimembranous | 0.2835 (0.0895)

4. Primary Outcome: Change in Muscle Function as Indicated by EMG Amplitude Assessed by Surface Electromyography (sEMG)
Description: as for outcome 3
Time Frame: week 9
Measure: Mean (Standard Deviation); unit: volts
Arm/Group | With C-brace
Number analyzed (Participants) | 11
volts
  Affected Tibialis anterior | 0.2639 (0.0897)
  Affected Soleus | 0.2776 (0.0755)
  Affected Medial gastrocnemius | 0.3312 (0.0950)
  Affected Vastus medialis | 0.2149 (0.1062)
  Affected Rectus femoris | 0.2146 (0.1072)
  Affected Biceps femoris | 0.2795 (0.0905)
  Affected Semimembranous | 0.2781 (0.1045)
  Unaffected Tibialis anterior | 0.3152 (0.0689)
  Unaffected Soleus | 0.3057 (0.0649)
  Unaffected Medial gastrocnemius | 0.2598 (0.0767)
  Unaffected Vastus medialis | 0.2770 (0.0812)
  Unaffected Rectus femoris | 0.2754 (0.0880)
  Unaffected Biceps femoris | 0.3026 (0.1161)
  Unaffected Semimembranous | 0.2877 (0.1002)

5. Primary Outcome: Metabolic Expenditure During Walking
Description: Change in metabolic expenditure during walking will be indicated by energy expenditure. Energy Expenditure will be measured by the K4 b2 Cosmed as follows: Oxygen cost will be calculated from oxygen consumption as the product of gait speed and body weight. Oxygen consumption will be collected on a breath-by-breath basis measured by a portable metabolic system (K4 b2 Cosmed). Prior to the testing, the system will be calibrated using room air and reference gas mixture. During the testing, the subject will wear a face mask and a heart rate monitor at all times and will be asked to breathe normally.
Time Frame: week 5
Population: Data were not collected for 2 participants.
Measure: Mean (Standard Deviation); unit: millilters/kilogram/minute (mL/kg/min)
Arm/Group | With C-brace
Number analyzed (Participants) | 12
millilters/kilogram/minute (mL/kg/min) | 0.03 (0.02)

6. Primary Outcome: Metabolic Expenditure During Walking
Description: as for outcome 5
Time Frame: week 9
Population: Data were not collected for 2 participants.
Measure: Mean (Standard Deviation); unit: millilters/kilogram/minute (mL/kg/min
Arm/Group | With C-brace
Number analyzed (Participants) | 12
millilters/kilogram/minute (mL/kg/min | 0.03 (0.01)

7. Secondary Outcome: Score on the Timed Up and Go Test
Description: Assesses mobility, balance, walking ability, and fall risk in older adults. The test measures the time it takes the subject to perform a sit to stand from a chair with arms, walk to a mark on the ground 10 feet away and return to the seated position in the chair with arms. This test has been used in assessing stroke recovery with high reliability and validity.
Time Frame: week 0
Population: Data were not collected for 3 participants.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | With C-brace
Number analyzed (Participants) | 11
seconds | 20.09 (12.38)

8. Secondary Outcome: Score on the Timed Up and Go Test
Description: as for outcome 7
Time Frame: week 5
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | With C-brace
Number analyzed (Participants) | 14
seconds | 19.37 (9.13)

9. Secondary Outcome: Score on the Timed Up and Go Test
Description: as for outcome 7
Time Frame: week 9
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | With C-brace
Number analyzed (Participants) | 14
seconds | 19.09 (9.75)

10. Secondary Outcome: Mental State as Assessed by the Folstein Mini Mental State Examination (MMSE)
Description: Mini Mental State Examination provides information about orientation, attention, learning, calculation, delayed recall, and construction. Several studies report acceptable validity of MMSE as a screening instrument and its relationship to functional outcome in stroke population. Total score ranges from 0 to 30, with a higher score indicating a better outcome.
Time Frame: week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | With C-brace
Number analyzed (Participants) | 14
score on a scale | 28.50 (2.14)

11. Secondary Outcome: Mental State as Assessed by the Folstein Mini Mental State Examination (MMSE)
Description: as for outcome 10
Time Frame: week 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | With C-brace
Number analyzed (Participants) | 14
score on a scale | 28.43 (2.65)

12. Secondary Outcome: Change in Hip Flexors Strength as Assessed by Dynamometry
Description: Muscle strength will be measured and quantified by using dynamometers on major bilateral lower limb muscles such as hip flexors.
Time Frame: week 0, week 9
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | With C-brace
Number analyzed (Participants) | 0

13. Secondary Outcome: Change in Hip Extensors Strength as Assessed by Dynamometry
Description: Muscle strength will be measured and quantified by using dynamometers on major bilateral lower limb muscles such as hip extensors.
Time Frame: week 0, week 9
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | With C-brace
Number analyzed (Participants) | 0

14. Secondary Outcome: Change in Hip Abductors Strength as Assessed by Dynamometry
Description: Muscle strength will be measured and quantified by using dynamometers on major bilateral lower limb muscles such as hip abductors.
Time Frame: week 0, week 9
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | With C-brace
Number analyzed (Participants) | 0

15. Secondary Outcome: Change in Hip Adductors Strength as Assessed by Dynamometry
Description: Muscle strength will be measured and quantified by using dynamometers on major bilateral lower limb muscles such as hip adductors.
Time Frame: week 0, week 9
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | With C-brace
Number analyzed (Participants) | 0

16. Secondary Outcome: Change in Knee Flexors Strength as Assessed by Dynamometry
Description: Muscle strength will be measured and quantified by using dynamometers on major bilateral lower limb muscles such as knee flexors.
Time Frame: week 0, week 9
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | With C-brace
Number analyzed (Participants) | 0

17. Secondary Outcome: Change in Knee Extensors Strength as Assessed by Dynamometry
Description: Muscle strength will be measured and quantified by using dynamometers on major bilateral lower limb muscles such as knee extensors.
Time Frame: week 0, week 9
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | With C-brace
Number analyzed (Participants) | 0

18. Secondary Outcome: Change in Ankle Dorsiflexors Strength as Assessed by Dynamometry
Description: Muscle strength will be measured and quantified by using dynamometers on major bilateral lower limb muscles such as ankle dorsiflexors.
Time Frame: week 0, week 9
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | With C-brace
Number analyzed (Participants) | 0

19. Secondary Outcome: Change in Ankle Plantarflexors. Strength as Assessed by Dynamometry
Description: Muscle strength will be measured and quantified by using dynamometers on major bilateral lower limb muscles such as ankle plantarflexors.
Time Frame: week 0, week 9
Population: Data for this outcome measure were not collected for any participant.
Arm/Group | With C-brace
Number analyzed (Participants) | 0

20. Secondary Outcome: Number of Participants With Bilateral Hip Range of Motion Within Normal Limits as Assessed by Goniometry
Description: Range of motion will be measured on bilateral hip using goniometry (goniometry is the use of a device called a goniometer to measure range of motion of a joint in degrees). After stroke, one side of the body is affected. For each participant, the range of motion of their affected hip will be measured and also the range of motion of their other hip (the unaffected hip) will be measured [it is possible that a participant will have a range of motion within normal limits on both hip sides (affected hip and unaffected hip)].
Time Frame: week 0
Measure: Count of Participants; unit: Participants
Arm/Group | With C-brace
Number analyzed (Participants) | 14
Participants
  Affected side hip flexion | 12
  Affected side hip extension | 11
  Affected side hip internal rotation | 13
  Affected side hip external rotation | 13
  Affected side hip abduction | 12
  Affected side hip adduction | 14
  Unaffected side hip flexion | 13
  Unaffected side hip extension | 13
  Unaffected side hip internal rotation | 13
  Unaffected side hip external rotation | 13
  Unaffected side hip abduction | 14
  Unaffected side hip adduction | 14

21. Secondary Outcome: Number of Participants With Bilateral Hip Range of Motion Within Normal Limits as Assessed by Goniometry
Description: as for outcome 20
Time Frame: week 9
Measure: Count of Participants; unit: Participants
Arm/Group | With C-brace
Number analyzed (Participants) | 14
Participants
  Affected side hip flexion | 13
  Affected side hip extension | 11
  Affected side hip internal rotation | 12
  Affected side hip external rotation | 11
  Affected side hip abduction | 13
  Affected side hip adduction | 14
  Unaffected side hip flexion | 14
  Unaffected side hip extension | 13
  Unaffected side hip internal rotation | 14
  Unaffected side hip external rotation | 14
  Unaffected side hip abduction | 14
  Unaffected side hip adduction | 14

22. Secondary Outcome: Number of Participants With Knee Joint Range of Motion Within Normal Limits as Assessed by Goniometry
Description: Range of motion will be measured on knee joints using goniometry (goniometry is the use of a device called a goniometer to measure range of motion of a joint in degrees). After stroke, one side of the body is affected. For each participant, the range of motion of their affected knee will be measured and also the range of motion of their other knee (the unaffected knee) will be measured [it is possible that a participant will have a range of motion within normal limits for both knees (affected knee and unaffected knee)].
Time Frame: week 0
Measure: Count of Participants; unit: Participants
Arm/Group | With C-brace
Number analyzed (Participants) | 14
Participants
  Affected side knee flexion | 11
  Affected side knee extension | 12
  Unaffected side knee flexion | 13
  Unaffected side knee extension | 12

23. Secondary Outcome: Number of Participants With Knee Joint Range of Motion Within Normal Limits as Assessed by Goniometry
Description: as for outcome 22
Time Frame: week 9
Measure: Count of Participants; unit: Participants
Arm/Group | With C-brace
Number analyzed (Participants) | 14
Participants
  Affected side knee flexion | 12
  Affected side knee extension | 14
  Unaffected side knee flexion | 14
  Unaffected side knee extension | 14

24. Secondary Outcome: Number of Participants With Ankle Joint Range of Motion Within Normal Limits as Assessed by Goniometry
Description: Range of motion will be measured on ankle joints using goniometry (goniometry is the use of a device called a goniometer to measure range of motion of a joint in degrees). After stroke, one side of the body is affected. For each participant, the range of motion of their affected ankle will be measured and also the range of motion of their other ankle (the unaffected ankle) will be measured [it is possible that a participant will have a range of motion within normal limits for both ankles (affected ankle and unaffected ankle)].
Time Frame: week 0
Measure: Count of Participants; unit: Participants
Arm/Group | With C-brace
Number analyzed (Participants) | 14
Participants
  Affected side ankle dorsiflexion | 4
  Affected side ankle plantarflexion | 13
  Unaffected side ankle dorsiflexion | 13
  Unaffected side ankle plantarflexion | 14

25. Secondary Outcome: Number of Participants With Ankle Joint Range of Motion Within Normal Limits as Assessed by Goniometry
Description: as for outcome 24
Time Frame: week 9
Measure: Count of Participants; unit: Participants
Arm/Group | With C-brace
Number analyzed (Participants) | 14
Participants
  Affected side ankle dorsiflexion | 6
  Affected side ankle plantarflexion | 12
  Unaffected side ankle dorsiflexion | 14
  Unaffected side ankle plantarflexion | 14

26. Secondary Outcome: Motor Impairment as Determined by the Fugl-Meyer Assessment
Description: The Fugl-Meyer Assessment evaluates and measures recovery of movement in individual post stroke. The Fugl-Meyer has been used in both clinical and research settings and is one of the most widely used quantitative measures of motor impairment. It uses an ordinal scale for scoring of 17 items for the lower limb component and 7 items on the balance component, for a total of 24 items. Each of the 24 items is scored as 0 (cannot perform), 1 (can perform partially), or 2 (can perform fully), with a total score ranging from 0 to 48, with a higher score indicating less impairment.
Time Frame: week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | With C-brace
Number analyzed (Participants) | 14
score on a scale | 23.43 (4.52)

27. Secondary Outcome: Motor Impairment as Determined by the Fugl-Meyer Assessment
Description: as for outcome 26
Time Frame: week 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | With C-brace
Number analyzed (Participants) | 14
score on a scale | 24.29 (5.27)

28. Secondary Outcome: Spasticity as Assessed by the Modified Ashworth Scale (MAS)
Description: This test measures spasticity in patients with lesions of the Central Nervous System by testing resistance to passive movement about a joint with varying degrees of velocity. Scores range from 0-4, with 0 indicating normal muscle tone and 4 indicating very high spasticity. The investigators will measure spasticity in lower limbs.
Time Frame: week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | With C-brace
Number analyzed (Participants) | 14
score on a scale
  Affected side hip flexor | 0 (0)
  Affected side hip extensor | 0.07 (0.27)
  Affected side knee flexors | 0.07 (0.27)
  Affected side knee extensors | 0.5 (0.76)
  Affected side ankle dorsiflexors | 0.21 (0.8)
  Affected side ankle plantarflexors | 0.71 (0.97)
  Unaffected side hip flexor | 0 (0)
  Unaffected side hip extensor | 0 (0)
  Unaffected side knee flexors | 0 (0)
  Unaffected side knee extensors | 0 (0)
  Unaffected side ankle dorsiflexors | 0 (0)
  Unaffected side ankle plantarflexors | 0 (0)

29. Secondary Outcome: Spasticity as Assessed by the Modified Ashworth Scale (MAS)
Description: as for outcome 28
Time Frame: week 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | With C-brace
Number analyzed (Participants) | 14
score on a scale
  Affected side hip flexor | 0.18 (0.46)
  Affected side hip extensor | 0.07 (0.27)
  Affected side knee flexors | 0.32 (0.54)
  Affected side knee extensors | 0.64 (0.72)
  Affected side ankle dorsiflexors | 0 (0)
  Affected side ankle plantarflexors | 0.57 (0.73)
  Unaffected side hip flexor | 0 (0)
  Unaffected side hip extensor | 0 (0)
  Unaffected side knee flexors | 0 (0)
  Unaffected side knee extensors | 0 (0)
  Unaffected side ankle dorsiflexors | 0 (0)
  Unaffected side ankle plantarflexors | 0 (0)

30. Secondary Outcome: Static Balance as Assessed by the Berg Balance Scale (BBS)
Description: A 14-item objective measure designed to assess static balance and fall risk in adult populations, with a total score range of 0 to 56 (higher scores represent better functional outcome). This test has been widely used to measure functional recovery in stroke patients with high reliability.
Time Frame: week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | With C-brace
Number analyzed (Participants) | 14
score on a scale | 48.64 (5.17)

31. Secondary Outcome: Static Balance as Assessed by the Berg Balance Scale (BBS)
Description: as for outcome 30
Time Frame: week 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | With C-brace
Number analyzed (Participants) | 14
score on a scale | 49.79 (4.51)

32. Secondary Outcome: Gait Speed as Assessed by the 10 Meter Walk Test (10MWT)
Description: Measure of gait speed. Subjects will walk a total of 14 meters at their preferred walking speed and at a fast pace. The test measures the time it takes the subject to complete the middle 10 meters of the walk.
Time Frame: week 0
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | With C-brace
Number analyzed (Participants) | 14
meters per second | 0.65 (0.28)

33. Secondary Outcome: Gait Speed as Assessed by the 10 Meter Walk Test (10MWT)
Description: as for outcome 32
Time Frame: week 5
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | With C-brace
Number analyzed (Participants) | 14
meters per second | 0.66 (0.31)

34. Secondary Outcome: Gait Speed as Assessed by the 10 Meter Walk Test (10MWT)
Description: as for outcome 32
Time Frame: week 9
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | With C-brace
Number analyzed (Participants) | 14
meters per second | 0.73 (0.29)

35. Secondary Outcome: Aerobic Capacity as Assessed by Peak VO₂ Per Kilogram Body Weight During the Six-minute Walk Test (6MWT)
Description: The participant will perform the 6MWT, in which the participant will walk as far as possible in six minutes. During the 6MWT, the peak volume of oxygen consumed per minute (peak VO₂) will be measured by a portable metabolic system. Data are reported as peak volume of oxygen (in milliliters) consumed per kilogram bodyweight per minute per meter walked [milliliters/kilogram/minute/meter (mL/kg/min/m)].
Time Frame: week 0
Measure: Mean (Standard Deviation); unit: mL/kg/min/m
Arm/Group | With C-brace
Number analyzed (Participants) | 14
mL/kg/min/m | 0.033 (0.015)

36. Secondary Outcome: Aerobic Capacity as Assessed by Peak VO₂ Per Kilogram Body Weight During the Six-minute Walk Test (6MWT)
Description: The participant will perform the 6MWT, in which the participant will walk as far as possible in six minutes. During the 6MWT, the peak volume of oxygen consumed per minute (peak VO₂) will be will be measured by a portable metabolic system. Data are reported as peak volume of oxygen (in milliliters) consumed per kilogram bodyweight per minute per meter walked [milliliters/kilogram/minute/meter (mL/kg/min/m)].
Time Frame: week 5
Population: Data for this outcome measure were not collected for 2 participants.
Measure: Mean (Standard Deviation); unit: mL/kg/min/m
Arm/Group | With C-brace
Number analyzed (Participants) | 12
mL/kg/min/m | 0.030 (0.015)

37. Secondary Outcome: Aerobic Capacity as Assessed by Peak VO₂ Per Kilogram Body Weight During the Six-minute Walk Test (6MWT)
Description: as for outcome 36
Time Frame: week 9
Measure: Mean (Standard Deviation); unit: mL/kg/min/m
Arm/Group | With C-brace
Number analyzed (Participants) | 14
mL/kg/min/m | 0.030 (0.013)

ADVERSE EVENTS:
Time Frame: 23 months
Description: 2 withdrew before adverse event data was collected.
Arm/Group | With C-brace
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 8/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | With C-brace (N=15)
Seizure (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | With C-brace (N=15)
Fall at home/office (General disorders) | 4 (4)
Skin pinch (Skin and subcutaneous tissue disorders) | 3 (5)
Blister (Skin and subcutaneous tissue disorders) | 1 (2)
Skin redness (Skin and subcutaneous tissue disorders) | 1 (1)
High blood pressure (General disorders) | 1 (1)
Device non-function (Investigations) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-16): https://cdn.clinicaltrials.gov/large-docs/60/NCT02892760/Prot_SAP_000.pdf